CLINICAL TRIAL: NCT05179291
Title: The Effects of Virtual Reality Glasses and External Cold and Vibration on Procedural Pain and Anxiety in Children During Venous Phlebotomy: Randomized Controlled Trial
Brief Title: Efficacy of VR and Buzzy on Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Diler Yilmaz, PhD, RN, Associate Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BANU-D-YILMAZ-002
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Procedural Pain; Procedural Anxiety; Pain; Children, Only
Keywords: Child; Child nursing; Non-pharmacological method; Pain relief
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buzzy Group (Experimental): In this group external cold and vibration-Buzzy was applied to the children during phlebotomy.
  Interventions: Other: Buzzy Group
- Virtual Realitiy-VR Group (Experimental): In this group Virtual Realitiy-VR was applied to the children during phlebotomy.
  Interventions: Other: Virtual Realitiy-VR Group
- Control Group (No Intervention): In this group, children received routine phlebotomy procedure

INTERVENTIONS:
Other: Buzzy Group — The Buzzy device was placed 5-10 cm above the injection area and making sure that it was in contact with the skin. The ice pack was kept in the deep freezer and placed into the device before the application. Buzzy was introduced to the children pre-procedure. Cold application and vibration were started pre-procedure and maintained until the procedure was completed. Following the Buzzy application, the device was wiped with 70% alcohol and used for other children. The Buzzy devices were kept in the deep freeze and refrozen. The same person conducted the pain reduction methods during phlebotomy.
  Arms: Buzzy Group
Other: Virtual Realitiy-VR Group — VR glasses were introduced to the children pre-procedure. The children were made to watch a video with VR glasses 2-3 minutes before starting the application and it continued until the end of the phlebotomy procedure (three minutes on average). 3D video suggestions (Space Experience, Blue Whale 360 VR Experience) were offered to the children before the phlebotomy procedure and they were asked to choose one of them.
  Arms: Virtual Realitiy-VR Group

SUMMARY:
The study was designed as a randomized controlled experimental research with the purpose of determining the effect of distraction by using external cold and vibration-Buzzy and VR on reducing procedural pain and anxiety in children aged 7 to 12 years during phlebotomy injection.

DETAILED DESCRIPTION:
In the literature, it is stated that nurses should use pharmacological and non-pharmacological methods in pain and anxiety management in painful procedures. Evidence-based studies are needed to show the effectiveness of non-pharmacological methods in reducing pain during invasive procedures and to investigate the effects of easy-to-apply methods on pain. In light of this information, this study aimed to compare the effect of distraction by using Buzzy and VR on reducing procedural pain and anxiety in children aged 7 to 12 years during phlebotomy.

This study is a prospective, randomized and controlled trial. Children aged 7 to 12 years who required phlebotomy were divided into three groups; buzzy, virtual reality, and controls. Data were obtained through face-to-face interviews with the children, their parents, and the observer before and after the procedure. The children's pain levels were assessed and reported by the parents and observers and the children themselves who self-reported using Wong-Baker FACES. The children's anxiety levels were also assessed using the Children's Fear Scale.

The study population consisted of children aged 7 to 12 years who presented to the children's phlebotomy room of the hospital.

Sample of the study consisted of a total of 120 children who met the sample selection criteria and were selected via randomization method.

Children were randomized into three groups: Buzzy (n= 40), VR group (n= 40), and the control group (n= 40).

Data were collected using the Information Form, Wong-Baker FACES Pain Rating Scale, Children's Fear Scale.

ELIGIBILITY:
Inclusion Criterial:

The sample selection criteria of the study were as follows: the children who

* were in the age group of 7-12 years,
* Due to undergo phlebotomy for blood testing,

Exclusion Criteria:

* had chronic diseases,
* had neuro-developmentally delayed,
* had visual, audio, or speech impairments,
* were hospital stay for treatment,
* had a history of sedative, analgesic or narcotic use within 24 hours before admission

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale | Through painful procedure completion, an average of 10 minutes
  In the study, pain level evaluations, the children's self-evaluations, parents' evaluations and the researcher's evaluations were carried out using the WB-FACES scale. This scale was developed by Donna Wong and Connie Morain Baker in 1988. The scale is graded between 0-10 points. A smiling face on the far left symbolizes "no pain" (0 very happy/no pain) and the pain increases from left to right. On the other hand, a crying face on the far right symbolizes "unbearable pain" (10 'hurts worst'). As the numbers increase in this scoring system, facial expressions also change referring to an increase in pain levels.
Children's Fear Scale | Through painful procedure completion, an average of 10 minutes
  CFS is used for measuring the child's anxiety level. CFS is a scale which makes an evaluation from 0 to 4 consisting of five facial expressions drawn to show expressions that vary from neutral expression (0=no anxiety) to scared face (4=severe anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University, Balıkesir, Bandirma, Turkey (Türkiye)